CLINICAL TRIAL: NCT01473797
Title: Evaluation of Efficacy and Tolerance of Cladribine in Symptomatic Patients With Pulmonary Langerhans Cell Histiocytosis and Impairment of Lung Function
Brief Title: Evaluation of Efficacy and Tolerance of Cladribine in Symptomatic Pulmonary Langerhans Cell Histiocytosis
Acronym: ECLA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOM10182; 2010-023344-32 (EudraCT Number)
Record Dates: First submitted 2011-10-14; First posted 2011-11-17 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Langerhans Cell Histiocytosis of Lung
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cladribine (Experimental)
  Interventions: Drug: Cladribine

INTERVENTIONS:
Drug: Cladribine — Subcutaneous injections, 0,1 mg/kg/day for 5 days, one course per month for 4 months

SUMMARY:
ECLA is a phase II, multicenter study testing sub cutaneous cladribine 0.1mg/kg/j during 5 days, administrated every month for 4 courses, in symptomatic adult patients with pulmonary Langerhans cell histiocytosis and impairment of lung function patients.

DETAILED DESCRIPTION:
ECLA is a phase II, multicenter study testing sub cutaneous cladribine 0.1mg/kg/j during 5 days, administrated every month for 4 courses, in symptomatic adult patients with pulmonary Langerhans cell histiocytosis and impairment of lung function patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 to 55 yr
* Histologically proven pulmonary Langerhans cell histiocytosis ( patients with presumptive diagnosis whose lung function precludes lung biopsy may be included after revision of their medical record at the national reference center for Langerhans cell histiocytosis)
* Symptomatic pulmonary Langerhans cell histiocytosis (NYHA dyspnea class ≥2) with:

  * irreversible airflow obstruction (FEV1/FVC<70%) with postbronchodilator FEV1 comprised between 30 and 70% of predicted
  * and/or decrease ≥15% in FEV1, FVC or DLCO as compared to baselines values in the year preceding the inclusion
* Signed written informed consent

Exclusion Criteria:

* Women at childbearing age without adequate contraception or wishing breastfeeding
* Male without adequate contraception during the study
* Dyspnea due to severe pulmonary arterial hypertension (PAP≥35mmHg) confirmed by cardiac right catheterism
* Previous malignancy
* Current infectious disease
* Renal failure
* Liver failure
* Severe alteration of lung
* Hematologic disease unrelated to Langerhans cell histiocytosis
* Epilepsy
* Hepatic, spleen or hematology involvement by Langerhans cell histiocytosis
* Pneumothorax within a month previously to inclusion
* Previous treatment with cladribine
* Contra indication to the use of cladribine
* Previous myelosuppressive treatment
* Simultaneous participation to another interventional clinical trial

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2018-04 (Actual); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Cumulated incidence of response to treatment | 6 months
  response to treatment after 6 months is defined as
  * ≥10% improvement of forced vital capacity (FVC)
  * and/or ≥10% improvement of postbronchodilator forced expiratory volume (FEV1) and ≥200ml

SECONDARY OUTCOMES:
Responses to treatment | 3 months
Absolute variations of FEV1, FVC, residual volume (RV), and Diffusing capacity of the lung for carbon monoxide (DLCO), (expressed in mL) | 6 months
Grade 3 or 4 neutropenia or thrombopenia | 6 months
Incidence of infection | 6 months
Incidence of grade 3 or 4 side effects | 6 months
Response to treatment of extra pulmonary localizations of the Langerhans disease | 6, 9, and 12 months
Incidence of pneumothorax | 12 months
Mortality | 12 months, 4 years
Incidence of secondary malignant disease | 4 years
Treatment response | at 6 months
Treatment response | 9 months
Treatment response | 12 months
Variation of nodular and cystic semiquantitative scores in High Resolution Computed Tomography (HRCT) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Abdellatif TAZI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Louis hospital, Paris, France

REFERENCES:
- [Derived] Benattia A, Lorillon G, de Margerie-Mellon C, Vercellino L, Bonniaud P, Marquette CH, Chevret S, Tazi A. Efficacy and safety of cladribine in adult pulmonary langerhans cell histiocytosis: a phase II study. Eur Respir J. 2026 Jan 29:2501464. doi: 10.1183/13993003.01464-2025. Online ahead of print. PMID 41611252